CLINICAL TRIAL: NCT02189668
Title: Non-operative Management of Uncomplicated Appendicitis With an Appendicolth in Children
Brief Title: Non-operative Management of Pediatric Appendicitis With an Appendicoltih
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High failure rate
Sponsor: Peter Minneci (Other)
Responsible Party: Sponsor-Investigator, Peter Minneci, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-00218
Record Dates: First submitted 2014-07-03; First posted 2014-07-14 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Appendicitis
Keywords: Appendicitis; Non-operative; Children; Appendicolith; fecalith; Pediatrics
MeSH Terms: conditions — Appendicitis; Fecal Impaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-operative Management (Experimental): Non-operative management with antibiotics only Zosyn (Piperacillin/Tazobactam) and then Augmentin unless penicillin allergic Cipro/Flagyl if penicillin allergic
  Interventions: Drug: Antibiotics only (Zosyn then Augmentin)
- Surgery (No Intervention): Usual care with urgent appendectomy

INTERVENTIONS:
Drug: Antibiotics only (Zosyn then Augmentin) — Intravenous and oral antibiotics without surgery Piperacillin/Tazobactam and then Augmentin Cipro/Flagyl if Penicillin allergic
  Other Names: non operative management
  Arms: Non-operative Management

SUMMARY:
To determine if non-operative management with antibiotics alone is a feasible treatment alternative for pediatric patients with uncomplicated acute appendicitis with an appendicolith identified on imaging.

DETAILED DESCRIPTION:
This study is a prospective randomized clinical trial comparing non-operative management with antibiotics to urgent appendectomy in children (ages 7-17yrs) with acute appendicitis with the presence of an appendicolith. Enrolled participants were followed up to 1 year post-discharge to observe the rates of appendicitis recurrence as well as identify the number of patients with complicated appendicitis as determined by pathologic examination.

ELIGIBILITY:
Inclusion Criteria:

* Age : 7-17 years
* Abdominal pain </= 48hours prior to receiving antibiotics
* White Blood Cell Count >5 but < 18
* US or CT confirmed early appendicitis plus:

  * US: </=1.1 cm in diameter, presence of appendicolith
  * CT: </= 1.1cm in diameter, presence of appendicolith

Exclusion Criteria:

* Positive urine pregnancy test
* Pain > 48 hours prior to first antibiotic dose
* Diffuse peritonitis
* History of chronic intermittent abdominal pain
* White Blood Cell count ≤ 5 or ≥ 18
* Absence of appendicolith or any evidence on imaging studies concerning for evolving perforated appendicitis including abscess or phlegmon

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Minneci, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minneci PC, Sulkowski JP, Nacion KM, Mahida JB, Cooper JN, Moss RL, Deans KJ. Feasibility of a nonoperative management strategy for uncomplicated acute appendicitis in children. J Am Coll Surg. 2014 Aug;219(2):272-9. doi: 10.1016/j.jamcollsurg.2014.02.031. Epub 2014 Apr 13. PMID 24951281
- [Result] Mahida JB, Lodwick DL, Nacion KM, Sulkowski JP, Leonhart KL, Cooper JN, Ambeba EJ, Deans KJ, Minneci PC. High failure rate of nonoperative management of acute appendicitis with an appendicolith in children. J Pediatr Surg. 2016 Jun;51(6):908-11. doi: 10.1016/j.jpedsurg.2016.02.056. Epub 2016 Mar 2. PMID 27018085

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-operative: Non-operative management with antibiotics alone Zosyn (Piperacillin/Tazobactam) and then Augmentin unless penicillin allergic Cipro/Flagyl if penicillin allergic
  Antibiotics only (Zosyn then Augmentin): Intravenous and oral antibiotics without surgery Piperacillin/Tazobactam and then Augmentin Cipro/Flagyl if Penicillin allergic
Period: Overall Study
Arm/Group | Non-operative | Surgery
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-operative | Surgery | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [13 to 14] | 11 [9 to 15] | 12 [11 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 5 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 2 | 8 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Did Not Have an Appendectomy
Description: Percentage of patients who were successfully managed nonoperatively with success defined as not undergoing appendectomy by one year after discharge
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Non-operative | Surgery
Number analyzed (Participants) | 5 | 9
Participants | 2 | 0

2. Secondary Outcome: Number of Participants With Complicated Appendicitis
Description: Percent of patients found to have complicated appendicitis (gangrenous or perforated) on pathologic examination.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Non-operative | Surgery
Number analyzed (Participants) | 5 | 9
Participants | 0 | 6

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for the duration of the follow-ups which was up to 1 year post-discharge.
Arm/Group | Non-operative | Surgery
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes